CLINICAL TRIAL: NCT04615819
Title: Access to Kidney Transplantation in Minority Populations (AKT-MP)
Brief Title: Access to Kidney Transplantation in Minority Populations
Acronym: AKT-MP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Case Western Reserve University (Other); University of Massachusetts, Amherst (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Larissa Myaskovsky, PhD, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-387 AKT-MP
Record Dates: First submitted 2020-08-07; First posted 2020-11-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Kidney Diseases
Keywords: Transplant
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): KTFT
  Interventions: Other: Kidney Transplant Fast Track (KTFT)
- Arm 2 (Experimental): PN
  Interventions: Other: Peer Navigation (PN)

INTERVENTIONS:
Other: Kidney Transplant Fast Track (KTFT) — Streamlined KT evaluation involving completion of most or all testing on the same day a patient arrives for their first pre-transplant clinic appointment. Or, a transplant clinic scheduler secures testing within a 4 week period.
  Arms: Arm 1
Other: Peer Navigation (PN) — Uses trained, previous KT recipients who meet weekly to monthly with patient participants to provide tailored information and assistance in completing the necessary steps to proceed to transplant.
  Arms: Arm 2

SUMMARY:
Hispanic/Latino (HL) and American Indian (AI) patients are more likely than whites to have kidney failure, but less likely to complete transplant evaluation or receive a kidney transplant (KT), the best treatment for kidney failure. Using comparative effectiveness research methods, we will conduct a pragmatic randomized trial to compare the efficacy and cost- effectiveness of two approaches to help HL and AI patients overcome barriers to completing transplant evaluation and receiving a KT: a streamlined KT evaluation process and a peer-assisted evaluation program; and, we will determine best practices to assist other transplant centers in implementing the better program. Findings from this work may help reduce disparities in transplant evaluation and KT.

DETAILED DESCRIPTION:
The AKT-MP study will assess whether Kidney Transplant Fast Track (KTFT), a streamlined KT evaluation process, or peer navigators (PN) who were former KT patients to help patients "navigate" their way through KT evaluation, can help vulnerable patients with kidney failure overcome barriers to transplant listing. After culturally and contextually adapting the two interventions, we will use a comparative effectiveness (CER) approach to conduct a pragmatic randomized trial of 398 kidney failure patients to compare the efficacy and effectiveness of the two approaches in disadvantaged groups at a university-affiliated transplant center with large HL and AI kidney failure patient populations, and we will compare results to historic comparison populations (local and national). We will assess facilitators and barriers to widespread implementation and conduct a cost effectiveness analysis. Although it is expected that KTFT will be more effective than PN, KTFT may also be more costly, requiring significant administrative and clinical changes in the transplant center, which may be impractical to maintain. Further, KTFT may lead to more patient ambivalence because the shortened evaluation period will give them less time to consider their treatment options. Thus, an important aspect of the proposed study is to comparative the effectiveness of the two methods. Ultimately, our study will inform transplant programs faced with disparities in KT about which disparity-reducing intervention to use given their particular needs and resources.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing kidney transplant evaluation at the University of New Mexico
* Greater than or equal to 18 years of age
* Mentally competent

Exclusion Criteria:

* Children less than 18 years of age are excluded because all research-related measurements are designed for patients over the age of 18. Children less than 18 years of age have dissimilar decision-making authority as a result of their developmental stage and dependency on adult guardians who must make all their transplant-related decisions, as required by all pediatric transplant centers. The proposed study focuses only on adult transplant patients.
* Waitlisted at another transplant center
* Prior kidney transplant
* Incarcerated patients
* Pregnant women
* Active systemic infection
* Non-skin malignancy or melanoma in the past 2 years
* Known cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of KT evaluation completion | Through study completion, an average of 1 year
  Completion of evaluation for KT and placement on the transplant waiting list.

SECONDARY OUTCOMES:
KT ambivalence | Through study completion, an average of 1 year
  KT ambivalence will be assessed with the Decisional Conflict Scale, with questions rating from strongly agree to strongly disagree.
Patient Reported Quality of Life | Through study completion, an average of 1 year
  We will use the PROMIS Scale v1.2 Global Health measure to assess quality of life (QOL), which includes items relevant to patients with kidney disease, including overall health, physical limitations, work, pain, energy, and emotional problems.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Myaskovsky, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT04615819/ICF_000.pdf